CLINICAL TRIAL: NCT02702232
Title: Shoulder Disorders in Patients With Parkinson's Disease
Status: Completed | Type: Observational
Sponsor: Shin Kong Wu Ho-Su Memorial Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: 20150802R; SKH-8302-105-DR-25 (Other Grant/Funding Number: Shin Kong Wu Ho-Su Memorial Hospital)
Record Dates: First submitted 2016-02-03; First posted 2016-03-08 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2018-01

CONDITIONS: Parkinson's Disease; Shoulder Pain
MeSH Terms: conditions — Parkinson Disease; Shoulder Pain | interventions — High-Energy Shock Waves

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Parkinson's disease: Patients with PD will be recruited consecutively from a neurology clinic. A group of sex- and age-matched normal subjects with be recruited from the public. These patients will be evaluated by ultrasonography for shoulder.
  Interventions: Other: Ultrasonography
- Normal: Normal controls who will be evaluated by ultrasonography for shoulder
  Interventions: Other: Ultrasonography

INTERVENTIONS:
Other: Ultrasonography — Ultrasonography is applied for normal subjects and patients with Parkinson's disease

SUMMARY:
Parkinson's disease (PD) is a multisystem neurodegenerative disorder that is increasingly recognized in our ageing population. It is characterized by cardinal clinical features including bradykinesia, tremor, rigidity, and postural instability. For most people with PD, the most serious concern is with the motor system: stiffness, slowness of movement, impaired handwriting and coordination, poor mobility and balance. However, more than half of all people with PD have experienced painful symptoms. Most people experience aching, stiffness, numbness and tingling at some point in the course of the illness. Defazio et al reported that pain may begin at clinical onset of PD or thereafter as a non-motor feature of PD.5 Aching muscles and joints are especially common in PD. Rigidity, lack of spontaneous movement, abnormalities of posture and awkward mechanical stresses all contribute to musculoskeletal pain in PD.

DETAILED DESCRIPTION:
One of the most common musculoskeletal complaints is shoulder pain or shoulder disorders, including frozen shoulder, bursitis, and rotator cuff lesions. Actually, shoulder pain or shoulder disorder can be the first sign of PD. The prevalence and severity of shoulder disorders in Parkinson's disease are not totally clear. In a retrospective study, Stamey found shoulder pain was present in 11% of patients with PD.

Over the past ten years ultrasound (US) has become popular in the evaluation of shoulder disorders. It allows for the detailed assessment of a wide range of changes involving different anatomic structures of the shoulder joint, including rotator cuffs, biceps tendon, and subdeltoid bursa. Koh et al found among 33 PD patients, 22 patients had abnormal US findings on the dominant side, and all 22 patients with abnormal US finding had a tendon tear and 9 patients had frozen shoulder. However, there were no control group in Koh' s study, and diagnosis of frozen shoulder with US findings is still controversial.

The purposes of this study are to evaluate patients with PD with a combination of physical examination and US study of the shoulder, and to compare the frequency and type of shoulder lesion in US between patients with PD and normal subjects. The investigators also plan to test the correlation between shoulder disorders or US abnormality and the severity of PD.

ELIGIBILITY:
Inclusion Criteria:

* Patients fulfilled the diagnosis of PD, as described by the United Kingdom Parkinson's Disease Society Brain Bank,
* Aged 50 to 80 years old.

Exclusion Criteria:

* Fracture or dislocation of the shoulder,
* Previous shoulder joint surgery,
* Severe medical comorbidities,
* Cognitive impairment (Mini-Mental Status Examination < 24).

Ages: 50 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with PD will be recruited consecutively from a neurology clinic. A group of sex- and age-matched normal subjects with be recruited from the public.
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2016-01; Primary Completion 2017-12 (Actual); Study Completion 2018-01 (Actual)

PRIMARY OUTCOMES:
Functional examination for diagnosis | 1 year
  The patient will received Cyriax's functional examination for shoulder joint to make a clinical diagnosis. It included three arm elevation, three tests for glenohumeral joints, and six resisted tests.
Ultrasound (US) examination for diagnosis | 1 year
  The patient will accept ultrasonography for shoulder joint for diagnosis

SECONDARY OUTCOMES:
Range of motion | 1 year
  The range of motion will showed in degrees. The range of motion measurement will include shoulder abduction, shoulder flexion, external rotation and internal rotation.
Pain | 1 year
  The VAS scores were obtained using a horizontal lines of 100 mm, with 0 on the left indicating no pain and 100 on the right indicating very severe pain. A VAS has been shown to be reliable and sensitive for quantifying pain, with test-retest reliability of >0.90.19 In previous studies of patients treated for various shoulder disorders, the responsiveness of VAS for pain was moderate to good.
Disability | 1 year
  The SPADI is a self-administered questionnaire to assess the pain and disability associated with shoulder disease. The total SPADI score is ranges between 0 and 100. The SDQ is a symptoms in patients with shoulder disorders. The final score is obtained by dividing the number by 100, which results in a final score ranging between 0 (no disability) and 100 (the worst situation).

CONTACTS AND LOCATIONS:
Locations (1):
- Shin Kong Wu Ho-Su Memorial Hospital, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hsieh LF, Kuo YC, Lin YT, Liu YF, Wang HC. Ultrasonographic imaging findings of the shoulder in patients with Parkinson disease. J Orthop Sci. 2023 Sep;28(5):1004-1010. doi: 10.1016/j.jos.2022.07.001. Epub 2022 Aug 6. PMID 35945122